CLINICAL TRIAL: NCT04208256
Title: The Neural Underpinnings of Disinhibited Eating Behavior in Adolescents With and Without Obesity
Brief Title: Food Intake and the Adolescent Brain
Acronym: ADOB
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-1171; K01DK120562 (NIH)
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Feeding Behavior; Brain; Adolescent
Keywords: pediatric obesity; resting-state functional magnetic resonance imaging; disinhibited eating behavior
MeSH Terms: conditions — Feeding Behavior; Pediatric Obesity | interventions — Aspartame; Glucola; Glucose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Energy Neutral: Bottled water (300 ml) with added fruit punch-flavored non-nutritive sweetener (aspartame) will be used as the energy neutral stimulus.
  Interventions: Dietary Supplement: Energy Stimulus
- Energy Surplus: 300ml fruit punch-flavored Glucola (75-gram[g], Azer Scientific) will be used as the energy surplus stimulus.
  Interventions: Dietary Supplement: Energy Stimulus

INTERVENTIONS:
Dietary Supplement: Energy Stimulus — Energy stimulus (energy surplus v. energy neutral) will be randomly assigned at the first brain imaging visit. At the second brain imaging visit, the participant will receive the alternate stimulus from what they received at the first brain imaging visit.
  Other Names: aspartame; Glucola; glucose

SUMMARY:
The brain plays an integral role in how and what people eat. However, the brain's contribution to overeating is not well understood during sensitive developmental periods such as adolescence, when excessive weight gain and obesity prevalence are a significant concern.The proposed study will use functional magnetic resonance imaging to examine how the brain's response to excess energy is related to overeating in adolescents with and without obesity.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* 13-18 years-old
* resident of Colorado

Exclusion Criteria:

* weigh less than 88 pounds or have a BMI% rank of <10% for age and sex;
* have a physician's diagnosis of metabolic syndrome or diabetes (Type 1 or 2);
* have a physician's diagnosis of anorexia nervosa or bulimia nervosa;
* currently taking anti-psychotic medications (not including anti-depressant or anti- anxiety medications);
* have a non-MRI safe device (e.g. pacemaker or defibrillator) or metal in the body (e.g. metal pins, shrapnel);
* experience symptoms of claustrophobia when in small or closed-off places;
* are pregnant or plan to become pregnant

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents with severe obesity enrolled from a specialty care lifesstyle medicine clinic and from the surrounding community. Adolescents with healthy weight enrolled from primary care clinic and from teh surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Brain function | brain imaging visit 1 (study visit 1); 30 minutes
  Brain function will be quantified via the blood oxygen level-dependent (BOLD) signal in the hypothalamus, insula, anterior cingulate cortex, nucleus accumbens, amygdala, and superior and inferior frontal gyri, and connectivity between these brain regions.
Disinhibited eating behavior | study visit 2; 1.5 hours
  Disinhibited eating behavior will be quantified via the kilocalories consumed during the test meal phase of the Eating in the Absence of Hunger laboratory protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No